CLINICAL TRIAL: NCT03297762
Title: Improving Adherence to Continuous Glucose Monitors in Publicly-insured Youth With Type 1 Diabetes
Brief Title: Increasing Use of Continuous Glucose Monitors in Publicly-insured Youth With Type 1 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment challenges
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Darrell M Wilson, Professor of Pediatrics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-36423
Record Dates: First submitted 2017-09-25; First posted 2017-09-29 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Type1diabetes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Gamification (Experimental): Use of continuous glucose monitor (Dexcom G5) with proactive intervention and incentives for time in use.
  Interventions: Behavioral: gamification; Behavioral: Use of Dexcom G5
- Standard care (Active Comparator): Use of continuous glucose monitor (Dexcom G5) per usual care.
  Interventions: Behavioral: Use of Dexcom G5

INTERVENTIONS:
Behavioral: gamification — incentives/rewards and contact between standard visits
  Arms: Gamification
Behavioral: Use of Dexcom G5 — Dexcom G5 continuous glucose monitor

SUMMARY:
To use an enhanced continuous glucose monitor (CGM) experience, including an automated CGM-electronic health record (EHR) data integration system, proactive interventions, and gamification techniques, to increase CGM use among publicly-insured youth with type 1 diabetes (T1D).

DETAILED DESCRIPTION:
The investigators will use an automated data integration system to monitor hours per week the CGM is worn and target interventions/troubleshooting techniques as needed. The investigators will use gamification techniques (i.e. ability to gain points and achieve small rewards) to help encourage CGM use and potentially improve glycemic control in this at-risk population.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes for more than 6 months
* on insulin pump or multiple daily injections without plans to change modality in next 6 months
* insured by CCS or Medi-Cal
* receiving care at Lucile Packard Children's Hospital or Stanford Children's Health outpatient clinics
* English or Spanish-speaking

Exclusion Criteria:

* major illness or condition that may alter glucose control or ability to complete the study including pregnancy, cystic fibrosis, cancer, liver disease, history of transplant, or hemoglobinopathy
* current oral glucocorticoid use
* prior use of a CGM system
* hemoglobin A1C <7.5% or >12%
* no wireless internet access

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
CGM use | baseline to 6 months
  amount of time per week CGM is used

SECONDARY OUTCOMES:
Hgb A1c | baseline to 6 months
  glycemic control as measured by Hgb A1c

CONTACTS AND LOCATIONS:
Overall Officials: Maria Chang, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Children's, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No